CLINICAL TRIAL: NCT03141320
Title: Confident Birthing: A Qualitative Study Exploring the Influences on Women's Confidence for Birth During Pregnancy and Labour
Brief Title: Confident Birthing: What Influences Women's Confidence for Birth?
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20007
Record Dates: First submitted 2017-03-14; First posted 2017-05-05 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy; Labour; Birth; Psychosocial Wellbeing; Woman's Health
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview/observation of social media comments — Interview with pregnant or postnatal women and observation of relevant social media comments

SUMMARY:
This is a grounded theory study aiming to understand women's perception of what influences their confidence for birth during labour and birth. Data is being collected using interviews and social media sources.

DETAILED DESCRIPTION:
This study aims to help women have a better birth experience, by trying to understand what a 'confident birth' means to women during pregnancy and labour. Results from a recent service evaluation at a local NHS Trust, exploring a new programme designed to enhance women's birth experience, highlighted the importance of understanding women's confidence for birth. A significant number of pregnant women that attended the course (19.5%) felt 'not at all confident' for birth. The service evaluation results also suggested that confidence for birth is an important influence of enhancing birth experience.

There is some research that suggests that if women's confidence for birth can be improved, then she may be less fearful of birth and have experience less labour pain. However, very little is known about what women consider to be a 'confident birth' and who or what they feel influences their confidence. If maternity services are able to understand this, this could possibly lead to the development of tools and strategies to help women to feel more confident for giving birth.

This is a qualitative study that involves two methods of data collection: interviews and social media. Women that are pregnant or have recently given birth will be interviewed to explore who or what they feel has influenced their confidence for birth. The interviews will last for about one and a half hours. The location for interview is flexible and women can be interviewed in their own home. In addition to this, approximately 500 messages posted on a large UK parenting website about confidence for birth will also be analysed.

ELIGIBILITY:
Inclusion Criteria:

* given birth within the last two years or are pregnant
* consider themselves well enough to take part in the study
* have received maternity care from specific NHS Trust

Exclusion Criteria:

* under 18 years old
* have not received maternity care from specific NHS Trust

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women or women that have given birth within the last two years
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Semi-structured interviews | 1 year

IPD SHARING:
Plan to Share IPD: No